CLINICAL TRIAL: NCT00998348
Title: Healthy Child Weight Through Improved Parent Practices and Environmental Change
Brief Title: Study of Parenting Intervention to Prevent Child Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dianne S. Ward, Faculty, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-0354; 1R01HL091093-01A1 (NIH)
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Obesity
Keywords: parenting; diet; physical activity; family; home; child
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comparison Group (No Intervention): The comparison group will receive children's picture books (1 per month for the duration of the 8-month program).
- Parenting Program (Experimental): The parenting program is an 8-month obesity prevention intervention for parents with preschool-age children.
  Interventions: Behavioral: Parenting Program

INTERVENTIONS:
Behavioral: Parenting Program — The parenting program is an 8-month intervention for parents with preschool-age children designed to teach strategies and skills that help parents better manage their day to day stresses of parenting while also promoting healthy lifestyle behaviors. Topics will include stress management, child management, family routines, emotion regulation, and coparenting. In later sessions parents will be encouraged to draw on these general parenting skills to promote healthier nutrition and physical practices at home. The intervention will be delivered through in-person group sessions (n=12) and tailored one-on-one telephone calls (n=11). A complementary child program will be delivered to children while parents are attending the group sessions.
  Other Names: Parenting SOS
  Arms: Parenting Program

SUMMARY:
This purpose of this project is to determine whether this 8-month parenting for healthy weight intervention is able to help parents improve their parenting skills and make positive changes in the nutrition and physical activity environment at home.

DETAILED DESCRIPTION:
The early years between ages 3-7 are critical in the development of obesity. The importance of the family in the development of children's eating and activity behaviors has been emphasized by experts, yet to date no obesity prevention interventions incorporating a strong family focus with emphasis on improved parenting practices have been developed. The work proposed here will address this gap by testing the efficacy of an 8-mo parenting intervention designed to change both social and physical aspects of the home environment, which in turn will reduced % body fat in children. Subjects will be 280 families (one parent and one child from each) with at least one preschool-age child (2-5 years old). Following baseline measures, pairs will be randomized into intervention or control. The intervention will teach more effective parenting skills (child management, communication, routines, etc.), then apply these skills to specific practices that encourage healthier behaviors. The intervention will include group sessions and tailored phone calls facilitated by a registered dietitian who has also received training in parent education. Group sessions will use multiple teaching strategies and include separate child activities. Tailored calls will use motivational interviewing techniques to help parents overcome barriers to behavior change. The intervention is guided by Darling and Steinberg's Integrative Model of parenting, which highlights the importance of parenting values, style and practices in child socialization, and Deci and Ryan's Self-Determination Theory, which suggests ways to foster autonomous motivation to adopt new behaviors. The resulting intervention will help parents learn skills to reduce their parenting-related stress and create home environments that support healthy-weight behaviors. The primary outcome, % body fat in children, will be assessed using anthropometry and a validated prediction equation (Dezenberg, 1999). Analyses will include baseline measurements of the outcome as a covariate. Secondary measures include child and parent diet and physical activity, parenting style and practices, and home environment. Maintenance effect will be assessed following a 6-mo no-intervention period. A comprehensive analysis is included to test for mediation effects. This intensive intervention will create the exposure necessary to make life-altering changes in weight-related behaviors. Plans build on extensive formative work conducted by our experienced researchers.

ELIGIBILITY:
Inclusion Criteria:

* Families must have at least one child age 2-5 years. The scientific rationale for focusing on this young population is that this age range includes the period often referred to as the "adiposity rebound," which has been identified as one of the critical periods for obesity development. Additionally, children of this age are still subject to strong parent and family influences which may be amenable to intervention.
* At least one parent or caregiver in the household must be overweight (BMI ≥25); however, this does not have to be the participating parent. The scientific rationale for focusing on families with at least one overweight parent is that having an overweight parent increases the child's risk of becoming overweight.
* Parents must be willing to participate in measures and intervention activities, and give consent for child's and his/her own participation.

Exclusion Criteria:

* Parents who are unable to speak English or comprehend standard age-level materials will be excluded. Currently funds are not available to translate and provide the program in Spanish or other languages.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Child percent body fat after the 8-month intervention period, controlling for baseline percent body fat. Percent body fat will be calculated using Dezenberg's equation which takes into account child height, weight, gender, race, and tricep skinfolds. | baseline, 8 months and 14 months

SECONDARY OUTCOMES:
Child BMI and Child BMI z-score based on measured child height, weight, and parent-reported date of birth | baseline, 8 months and 14 months
Parent BMI based on measured height and weight | baseline, 8 months and 14 months
Parent and child dietary intake measured with 3 unannounced dietary recalls collected via telephone interview (will not include foods eaten by child while outside of parent's care) | baseline, 8 months and 14 months
Parent and child physical activities assessed via 7-days of accelerometer monitoring (using the AciGraph GT3X monitor programed with 60-s epochs for adults and 15-s epochs for children) | baseline, 8 months and 14 months
Parenting-related stress assessed with the Parental Stress Index - Short Form (Abidin, 1995) | baseline, 8 months and 14 months
Autonomous motivation to change behaviors (parenting practices, feeding practices, and physical activity practices) will be assessed using modified versions of the Treatment Self-Regulation Questionnaire (Williams GC, 1996) | baseline, 8 months and 14 months
Self-efficacy for general parenting will be assessed with the Parenting Sense of Competence Scale (Johnston C, 1989) | baseline, 8 months and 14 months
Self-efficacy for implementing healthy nutrition and physical activity practices will be assessed with an instrument recently developed by the PI. | baseline, 8 months and 14 months
Parents' perceived social support and connectedness with regard to positive parenting and healthy feeding and physical activity practices will be assessed using modified versions of the Social Provisions Scale (Cutrona, 1987) | baseline, 8 months and 14 months
The Alabama Parenting Questionnaire - Preschool Revision (Clerkin, 2007)will be used to assess general parenting practices, specifically the use of positive parenting, inconsistent parenting, and punitive parenting | baseline, 8 months and 14 months
Difficulties in Emotion Regulation (Gratz, 2004) will be used to assess parental skills at regulating their own emotions | baseline, 8 months and 14 months
Coping with Children's Negative Emotions (Fabes, 1990) will be used to assess parental skill at helping the child deal with and manage his/her negative emotions | baseline, 8 months and 14 months
Confusion, Hubbub, and Order Scale (Matheny, 1995) will be used to assess the degree of order versus confusion in the home environment | baseline, 8 months and 14 months
The Parenting Convergence Scale (Ahrons, 1981) will be used to assess parental skill with coparenting | baseline, 8 months and 14 months
The Caregiver Feeding Style Questionnaire (Hughes SO, 2005) will be used to assess the two dimensions of parenting: demandingness and responsiveness as they relate to feeding practices | baseline, 8 months and 14 months
The Parental Feeding Style Questionnaire (Wardle, 2002) will be used to assess parents' use of emotional feeding, instrumental feeding, encouraging to eat, and control over eating | baseline, 8 months and 14 months
Nine subscales from the Comprehensive Feeding Practices Questionnaire (Musher-Eizenman, 2007) will be used to assess child control, encouraging balance/variety, involvement, modeling, monitoring, pressure to eat, restriction for health or weight control, | baseline, 8 months and 14 months
One sub-scale from the Preschooler Feeding Questionnaire (Baughcum, 2001) will be used to assess structure during feeding interactions | baseline, 8 months and 14 months
Two items slightly modified from the Child Feeding Questionnaire (Birch, 2001) will be used to determine parent perceptions of child weight and concern about child becoming overweight | baseline, 8 months and 14 months
A variety of newly developed items drawn from the literature will be used to assess parent practices around child physical activity | baseline, 8 months and 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Dianne S Ward, EdD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Health Promotion and Disease Prevention, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ward DS, Vaughn AE, Bangdiwala KI, Campbell M, Jones DJ, Panter AT, Stevens J. Integrating a family-focused approach into child obesity prevention: rationale and design for the My Parenting SOS study randomized control trial. BMC Public Health. 2011 Jun 5;11:431. doi: 10.1186/1471-2458-11-431. PMID 21639940